CLINICAL TRIAL: NCT01098721
Title: A Double-blinded, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Topically Applied 1.0% WBI-1001 Cream for 12 Weeks, in the Treatment of Mild to Moderate Plaque Psoriasis.
Brief Title: A Safety/Efficacy Study of a Non-steroid, Topical Cream Treatment of Psoriasis Over 12-weeks
Acronym: 134993
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Welichem Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WBI-1001-102; 134993 (Registry Identifier: Health Canada, Therapeutic Products Directorate)
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Psoriasis
Keywords: plaque psoriasis; skin diseases; anti-inflammatory; non-steroid; topical cream
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — tapinarof

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Placebo Comparator): A placebo cream applied topically twice daily (BID)by each of 20 patients, once in the morning and once in the evening for 12 weeks.
  Interventions: Drug: WBI-1001
- Group 2 (Active Comparator): A 1.0% WBI-1001 cream applied topically twice daily (BID) by each of 40 patients, once in the morning and once in the evening for 12 weeks.
  Interventions: Drug: WBI-1001

INTERVENTIONS:
Drug: WBI-1001 — Comparison of two doses (0% and 1.0%) of the the WBI-1001 cream applied topically, twice daily for 12 weeks.

SUMMARY:
Psoriasis is a chronic inflammatory skin disorder that is characterized by hyperproliferation of the keratinocytes and inflammation of the epidermal and dermal layers of the skin. This study, in patients with mild to moderate plaque psoriasis, is designed to further determine the efficacy, safety and tolerability of the novel, topically applied, non-steroid, anti-inflammatory WBI-1001 cream over a period of 12 weeks.

DETAILED DESCRIPTION:
A double-blinded, placebo-controlled study. Following screening, eligible patients will be randomized on Day 0 into one of two treatment groups in a 1:2 ratio:

Group 1: placebo (vehicle) cream, twice daily (BID). Group 2: 1.0% WBI-1001 cream, BID. Patients will be randomized to treat all treatable lesion areas except for the face, scalp, groin and genital areas, and will be instructed to apply the cream twice daily for 84 days, at the same time each day, once in the morning and once in the evening.

During the study patients will visit the study centre for assessment of efficacy, safety and tolerability at 0, 14, 28, 56 and 84 days after initiation, and patients will be phoned at Day 112 for a follow-up safety assessment.

Patients that withdraw from the study before Day 56 due to reasons other than adverse events will be replaced as necessary to ensure that there are at least 16 patients from the placebo and 32 from the active cream treated groups remaining in the study at Day 56.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of stable plaque psoriasis for at least 6 months representing a maximum of 10% of BSA with a minimum of 1% BSA excluding the face, groin ,scalp and genital regions and with a minimum of one target plaque that is at least 2 x 2 cm in size at Day 0.
* PGA of 2 to 4 at Day 0.
* In good general health and free of any disease state or physical condition that might impair the evaluation of plaque psoriasis.
* Women of child bearing potential (WOCBP) must have a negative serum beta-human chorionic gonadotrophin (b-hCG) pregnancy test before randomization. WOBCP who are not abstinent from sex with male partners may be entered into the study if they are willing to continue to use adequate contraceptive precautions for the duration of the study. Male patients with female sexual partners who are able to become pregnant must ensure that an acceptable method of birth control is used while they are in the study. Women who are lactating will not be eligible for the study.
* Willing and able to comply with the protocol and likely to attend all study visits.
* Provide written, informed consent prior to the initiation of any study-related procedures.

Exclusion Criteria:

* Spontaneously improving or rapidly deteriorating plaque psoriasis.
* Any other skin diseases that might interfere with the clinical assessment of plaque psoriasis and/or put the patient at risk.
* Pustular, erythrodermic or other non-plaque forms pf psoriasis.
* Guttate psoriasis as the dominant form of psoriasis.
* Other concomitant, serious illness or medical condition (eg., human immunodeficiency virus, renal insufficiency, clinically significant abnormal laboratory values) that could put the patient at risk during the study.
* History of neurological/psychiatric disorders, including psychotic disorders or dementia, or any other reason that would interfere with the patient's participation in the trial.
* Systemic immunomodulatory therapy known to affect psoriasis and decreases immune cell populations (eg., alefacept) within 24 weeks of the baseline visit.
* Systemic immunomodulatory therapy known to affect psoriasis and that does not typically decrease immune cell populations (eg., etanercept) within 12 weeks prior to the baseline visit.
* Any phototherapy (including laser for the treatment of psoriasis), photo-chemotherapy,or systemic psoriasis therapy (such as systemic corticosteroids, methotrexate, retinoids or cyclosporine) within 4 weeks prior to the baseline visit.
* Prolonged exposure to artificial or natural sources of ultraviolet radiation within 4 weeks prior to the baseline visit or intention to have such exposure during the study, thought by the investigator likely to modify the patient's psoriasis.
* Topical anti-psoriatic therapy (including topical retinoids and vitamin D analogs) on the areas to be treated within 2 weeks prior to the baseline visit.
* Alcohol abuse during the last 2 years as defined by the consumption of >14 standard drinks of alcohol per week.
* Use of lithium within 2 weeks prior to the screening visit.
* Use of beta blockers (eg., propranolol) within 2 weeks prior to the screening visit unless on a stable dose for >3 months.
* Known or suspected hypersensitivity to any of the constituents of the investigational product.
* Treatment with an investigational drug within 1 month of Day 0 or current participation in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Day 0) in PGA in patients randomized to placebo as compared to patients randomized to 1.0% WBI-1001. | 84 days
  The primary indication of efficacy will be demonstrated by improvement in the Physician's Global Assessment (PGA) in patients treated with the active (1.0% WBI-1001) cream as compared with those treated with the placebo cream.

SECONDARY OUTCOMES:
Change in PASI score from baseline (Day 0) to Day 84 for patients in Group 1 compared with those in Group 2. | 84 days
  Change in the Psoriasis Area and Severity Index (PASI) score from the baseline (Day 0) at Day 84 in patients randomized to the placebo compared with those randomized to the 1.0% WBI-1001 cream treatment.
Blood and urine analyses and vital signs assessments of patients from Day 0 to Day 84, and the follow-up at Day 112. | 84 days plus 112 day follow-up.
  Comparative assessment of the laboratory analyses and vital signs of Group 1 and Group 2 patients from Day 0 to Day 84, and the follow-up at Day 112.
Change from baseline in BSA at Day 84 in patients randomized to placebo compared with those randomized to 1.0% WBI-1001 cream treatment. | 84 days
  Change in the BSA of involved skin (except for the face, scalp, groin and genital areas) from that at baseline (Day 0) to that at Day 84 when comparing patients in Group 1 with those in Group 2.
Change from baseline (Day 0) in mean target lesion score at Day 84 in patients in Group 1 compared with those in Group 2. | 84 days
Change from baseline (Day 0)in target lesion induration at Day 84 in patients in Group 1 compared with those in Group 2. | 84 days
Change from baseline (Day 0) in target lesion scaling at Day 84 in patients in Group 1 compared with those in Group 2. | 84 days
Change from baseline (Day 0)in target lesion erythema at Day 84 in patients from Group 1 compared with those from Group 2. | 84 days
Type, frequency, severity and relationship of adverse events in patients from Group 1 compared with those from Group 2. | 84 days + follow-up at 112 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, MSc, Principal Investigator — Innovaderm Research Inc.